CLINICAL TRIAL: NCT06955624
Title: Use of Omics Methods to Classify Variations of Uncertain Significance and Improve Diagnosis of Neurogenetic Diseases
Acronym: OMID-NEURO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Collaborators: University Hospital, Lille (Other); Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024/0190/HP; 2024-A01559-38 (Registry Identifier: RCB)
Record Dates: First submitted 2025-04-15; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Neurogenetic Diseases
Keywords: Neurogenetic diseases; Central nervous system disease
MeSH Terms: conditions — Central Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Qualification: Category 2 Product or procedure: excluding health products (products not mentioned in Article L.5311-11 of the Public Health Code)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Controls (Other): * Patients with neurological disease affecting the central nervous system, of confirmed monogenic or probable oligogenic cause (positive controls
  * Unaffected relatives, showing no symptoms of the disease after the expected age of onset of symptoms in the family
  Interventions: Genetic: RNA and/or DNA methylation and/or protein analysis

INTERVENTIONS:
Genetic: RNA and/or DNA methylation and/or protein analysis — RNA and/or DNA methylation and/or protein analysis from a blood sample or another tissue including dedifferenciation into induced pluripotent stem cells

SUMMARY:
Many neurological disorders show a strong genetic basis, from hereditary diseases caused by a single mutation in a given gene, to diseases caused by combinations of strong genetic risk factors. However, even after the sequencing of the appropriate genes, a large proportion of patients remains undiagnosed, either because there is no candidate mutation observed, or in case of identification of a candidate mutation with insufficient knowledge to consider it as pathogenic or not.

The aim of this project is to identify the cause of neurogenetic diseases in patients in situations of diagnostic wandering or dead ends by proposing the analysis of RNA and/or proteins from different tissues.

ELIGIBILITY:
Inclusion Criteria:

For this project, the inclusion of 3 participant profiles is required:

* 1a. Patient, major or minor, with a neurological disease affecting the central nervous system, who has already benefited from a genomic analysis (panel, exome or genome sequencing) as part of routine care, with inconclusive analysis because the result was either a variation of uncertain significance or the absence of a variant of interest (patients with inconclusive genomic results).
* 1b. Patient with neurological disease affecting the central nervous system, of confirmed monogenic or probable oligogenic cause (positive controls).
* A relative of a type 1a. or 1b. patient with no symptoms of the disease, after the expected age of onset of symptoms in the patient's own family (healthy relatives).

For all 3 groups:

* Affiliation with a social security scheme
* Agreement to take part in the study with signature of a specific informed consent form for the study.

Exclusion Criteria:

For patients with inconclusive results: Patient with a neurological disease not suspected of a monogenic or oligogenic cause

For healthy relatives: existence of a neurological disease (other than uncomplicated migraine) or psychiatric disease (other than simple anxiety stable under treatment).

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2030-01-15 (Estimated); Study Completion 2031-01-15 (Estimated)

PRIMARY OUTCOMES:
number and proportion of patients | through study completion, an average of 5 years
  number and proportion of patients in the "Patients with inconclusive results" group for whom a final diagnosis can be made at the end of this research.

SECONDARY OUTCOMES:
Inclusion | through study completion, an average of 5 years
  Inclusion of at least 50 participants with successful implementation of at least two procedures (see below, list of procedures)
Identification of at least one candidate biomarker linked to one or more abnormalities of a gene or group of genes. | through study completion, an average of 5 years
  Identification of at least one candidate biomarker linked to one or more abnormalities of a gene or group of genes.

CONTACTS AND LOCATIONS:
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No